CLINICAL TRIAL: NCT01937247
Title: Redesigned Process in the Operating Room: Monitoring and Evaluating Success of Reducing Non Operative Time
Brief Title: Redesigned Process in the Operating Room
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Roland Kaddoum, Assistant Professor, MD, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ANES.RK.04; AUBMC (Other: AUBMC)
Record Dates: First submitted 2013-08-29; First posted 2013-09-09 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Non-operative Time; General Surgery, Above 18 Years of Age
Keywords: Operative Time; Operating Rooms; Efficiency
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard process (Placebo Comparator): The control group is placebo group and this is our standard practice. Patients will be induced in the operating room and at the end of surgery will be reversed with neostigmine 50µg/kg and glycopyrrolate 10µg/kg. Once extubated and rolled out of the room, the house keeper team will start cleaning the operating room
  Interventions: Procedure: STANDARD PROCESS
- Redesigned process (Active Comparator): Patients will be inducted in the induction room. At the end of surgery and after placement of the surgical dressing, the registered nurse will call in the house keeper to start cleaning of the OR (parallel processing) before the patient exits the room. The patient will be reversed with sugammadex 4mg/kg IV
  Interventions: Procedure: Patients will be inducted in the induction room; Procedure: Redesigned process; Drug: patient will be reversed with sugammadex 4mg/kg IV

INTERVENTIONS:
Procedure: Patients will be inducted in the induction room — The patients will be inducted in the induction room
  Arms: Redesigned process
Procedure: Redesigned process — The registered nurse will call in the house keeper to start cleaning of the OR (parallel processing) before the patient exits the room
  Arms: Redesigned process
Drug: patient will be reversed with sugammadex 4mg/kg IV — The patient will be reversed with sugammadex 4mg/kg IV, and then extubated before being moved out of the OR
  Arms: Redesigned process
Procedure: STANDARD PROCESS — standard process
  Arms: Standard process

SUMMARY:
The main purpose of the study is to examine whether operating room (OR) efficiency will be improved by significantly decreasing non operative time. This study also aims: 1) to evaluate whether a decrease in non-operative time will result in increased surgeon and staff satisfaction, 2) to determine whether there is an increase in the complication rate during the redesigned process perioperatively and until discharge from the post anesthesia care unit, and 3) to rate patient satisfaction.

DETAILED DESCRIPTION:
The study aims to examine whether operating room efficiency will be improved by decreasing non operative time while ensuring patient safety.

Patients will be randomized into one of two groups:

In group A (new process): patients will be inducted in the induction room. At the end of surgery and after placement of the surgical dressing, the registered nurse will call in the house keeper to start cleaning of the OR (parallel processing) before the patient exits the room. The patient will be reversed with sugammadex 4mg/kg IV, and then extubated before being moved out of the OR. In group B (the current practice at AUBMC), patients will be treated as follows: patients will be induced in the operating room and at the end of surgery will be reversed with neostigmine 50µg/kg and glycopyrrolate 10µg/kg. Once extubated and rolled out of the room, the house keeper team will start cleaning the operating room. Induction time (IT), emergence time (ET), and turn over time (TOT) will be recorded for both groups.

We expect to show that OR efficiency will be improved by significantly decreasing non operative time while ensuring patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients, above 18 years of age, undergoing general surgery for surgeon X under general anesthesia
* Patients undergoing only the following general surgeries: laparoscopic hernia, laparoscopic appendectomy, laparoscopic cholecystectomy, and laparoscopic gastric/band sleeve surgeries
* American Society of Anesthesiologist Physical Status (ASA) I or II
* Research participant willing to sign informed written consent.

Exclusion Criteria:

* Patients under 18 years of age
* Patients undergoing general surgery for surgeon X under regional or spinal anesthesia
* Patients undergoing surgeries other than the following: laparoscopic hernia, laparoscopic appendectomy, laparoscopic cholecystectomy, and laparoscopic gastric/band sleeve surgeries
* American Society of Anesthesiologist Physical Status (ASA) III, IV, V, and VI
* Emergency and lifesaving Cases
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Inability to bring the next patient to the induction room for uncontrollable reasons such as failure of equipment, late arrival to the hospital, or late financial or medical clearance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Non-operative time | within 24 hours of surgery
  For Group A, non-operative time is defined as induction, emergence and turnover time For Group B, non-operative time is defined as turnover time

SECONDARY OUTCOMES:
Satisfaction of the operation room staff and surgeons with the redesigned process | within 24-48 hours after surgery
  semi-structured individual interviews
Patient satisfaction | within 24-48 hours aftery surgery
  Patient satisfaction survey
Complication rate | wihtin 24 hours of srugery

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kaddoum, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaddoum R, Tarraf S, Shebbo FM, Bou Ali A, Karam C, Abi Shadid C, Bouez J, Aouad MT. Reduction of Nonoperative Time Using the Induction Room, Parallel Processing, and Sugammadex: A Randomized Clinical Trial. Anesth Analg. 2022 Aug 1;135(2):406-413. doi: 10.1213/ANE.0000000000006102. Epub 2022 Jun 3. PMID 35839499